CLINICAL TRIAL: NCT07185490
Title: Exploratory Clinical Study Protocol on the Safety and Efficacy of Fully Human BCMA-Targeted Chimeric Antigen Receptor Autologous T-Cell Injection (IASO104) for the Treatment of Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: IASO104 for the Treatment of Patients With Relapsed/Refractory Multiple Myeloma
Acronym: IASO104
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025081; Nanjing Reindeer Biotechnology (Other Grant/Funding Number: Nanjing Reindeer Biotechnology Co., Ltd.)
Record Dates: First submitted 2025-09-05; First posted 2025-09-22 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-11

CONDITIONS: Relapsed/Refractory Multiple Myeloma (RRMM); Plasma Cell Leukemia (PCL)
MeSH Terms: conditions — Multiple Myeloma; Leukemia, Plasma Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IASO104 (Experimental): IASO104 will be administered in one infusion.
  Interventions: Biological: IASO104

INTERVENTIONS:
Biological: IASO104 — IASO104 is a personalized, BCMA-targeted, genetically modified autologous T-cell immunotherapy product.

SUMMARY:
This study is a single-center, open-label, dose-exploration trial designed to evaluate the tolerability and safety of different doses of IASO104 in patients with relapsed/refractory plasma cell neoplasms, determine the recommended dose of IASO104, and assess its pharmacokinetic and pharmacodynamic characteristics. Additionally, the study will preliminarily observe the efficacy of the investigational drug in a small sample of subjects with relapsed/refractory multiple myeloma.

DETAILED DESCRIPTION:
This study adopts a "3+3" dose-escalation design, with three predefined dose levels: 0.5×10⁶ CAR-T cells/kg, 1.0×10⁶ CAR-T cells/kg, and 3.0×10⁶ CAR-T cells/kg, administered as a single infusion.For each dose group, the first subject must be observed for at least 2 weeks after infusion before subsequent subjects can be treated. If stable biological activity or clinical benefit is observed at a lower dose level, the study may proceed with 1-2 expanded dose groups at lower levels after discussion between the investigator and sponsor, without requiring MTD determination.During the dose-escalation phase, 2-3 subjects will be enrolled per dose level, with the total number of subjects depending on the escalation progression (estimated 4-6 subjects in this phase). Treatment in the next dose group may only begin after all subjects in the current group have completed DLT assessment post-infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years, any gender.
2. Diagnosis of multiple myeloma (MM) per International Myeloma Working Group (IMWG) diagnostic criteria.
3. Prior therapy requirements:

   MM patients: ≥3 prior lines of therapy, including:
   * 1 proteasome inhibitor (PI)
   * 1 immunomodulatory drug (IMiD)
   * 1 anti-CD38 monoclonal antibody Exception: No minimum line requirement for subjects refractory to PIs, IMiDs, and anti-CD38 therapy.

   Primary plasma cell leukemia (pPCL): ≥1 prior line including ≥1 PI and ≥1 IMiD.
4. Documented disease progression during/within 12 months after last anti-myeloma therapy (exemption: No 12-month requirement if last line was CAR-T).
5. Measurable disease at screening (≥1 of the following):

   Serum M-protein:

   IgG ≥10 g/L IgA/IgD/IgE/IgM ≥5 g/L Urine M-protein ≥200 mg/24h Serum free light chains (FLC): Involved FLC ≥100 mg/L with abnormal κ/λ ratio Bone marrow plasma cells ≥30% (if no measurable M-protein/FLC).
6. ECOG performance status 0-1.
7. Life expectancy ≥12 weeks.
8. Adequate organ function (all lab values within 7 days prior to enrollment):

   Hematology:

   Absolute neutrophil count (ANC) ≥1×10⁹/L (allowed: growth factor support, but none within 7 days) Absolute lymphocyte count (ALC) ≥0.3×10⁹/L Platelets ≥50×10⁹/L (no transfusion within 7 days) Hemoglobin ≥60 g/L (no RBC transfusion within 7 days; erythropoietin allowed)

   Liver:

   ALT/AST ≤2.5×ULN Total bilirubin ≤1.5×ULN Renal: Calculated CrCl ≥40 mL/min (Cockcroft-Gault)

   Coagulation:

   Fibrinogen ≥1.0 g/L aPTT/PT ≤1.5×ULN Pulmonary: SpO₂ >91% (room air) Cardiac: LVEF ≥50% (echocardiography).
9. Contraception: Subjects/partners must use effective contraception from consent through 1 year post CAR-T infusion (excluded: calendar method).
10. Signed informed consent approved by the Ethics Committee prior to screening.

Exclusion Criteria:

1. Active graft-versus-host disease (GVHD) or requiring long-term immunosuppressive therapy.
2. Prior hematopoietic stem cell transplantation (HSCT):

   Autologous HSCT (Auto-HSCT) within 12 weeks before apheresis,

   ≥2 prior Auto-HSCTs, Any prior allogeneic HSCT (Allo-HSCT).
3. Prior cell therapy targeting plasma cells within 3 months before apheresis, or detectable residual cellular therapy products in peripheral blood.
4. Recent anti-myeloma therapies (relative to apheresis):

   Monoclonal antibody treatment within 21 days, Cytotoxic chemotherapy or proteasome inhibitors within 14 days, Immunomodulatory drugs within 7 days, Other anti-tumor therapies within 14 days or 5 half-lives (whichever is shorter).
5. Chronic corticosteroid use (>20 mg/day prednisone or equivalent), except for physiologic replacement, topical, or inhaled use.
6. Uncontrolled hypertension despite medication.
7. Severe cardiac disease, including:

   Unstable angina, Myocardial infarction (within 6 months before screening), Congestive heart failure (NYHA Class ≥III), Severe arrhythmias.
8. Unstable systemic illnesses per investigator's judgment (e.g., severe hepatic, renal, or metabolic disorders requiring medication).
9. Other malignancies within 5 years, excluding:

   Carcinoma in situ of the cervix, Basal/squamous cell skin cancer, Localized prostate cancer post-radical resection, Ductal breast carcinoma in situ post-resection.
10. History of solid organ transplantation.
11. Suspected or confirmed CNS involvement by plasma cell neoplasms.
12. Major surgery within 2 weeks before apheresis or planned within 2 weeks post-treatment (allowed: minor procedures under local anesthesia).
13. Investigational drugs within 1 month before apheresis.
14. Uncontrolled active infections:

    Persistent symptoms despite appropriate therapy, Requiring IV antimicrobials at screening.
15. Viral infections:

    HBV: HBsAg(+) or HBcAb(+) with detectable HBV DNA, HCV: HCV Ab(+) with detectable HCV RNA, HIV Ab(+), CMV DNA(+), Syphilis: TRUST(+) and TPPA(+).
16. Pregnancy or lactation.
17. Psychiatric disorders, cognitive impairment, or active CNS diseases.
18. Other conditions deemed ineligible by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-08-15 (Estimated); Study Completion 2029-08-15 (Estimated)

PRIMARY OUTCOMES:
incidence and severity of adverse events (AEs) | Minimum 2 years after IASO104 infusion

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Minimum 2 years after IASO104 infusion
  The proportion of subjects achieving stringent complete response (sCR), complete response (CR), very good partial response (VGPR), and partial response (PR) after treatment with IASO104 injection
Duration of Response (DOR) | Minimum 2 years after IASO104 infusion
  Duration of response (DOR) was defined as the time from the first documented achievement of response (≥ partial response [PR]) to disease progression or death from any cause (whichever occurred first) in subjects treated with IASO104 injection.
Progression-Free Survival (PFS) | Minimum 2 years after IASO104 infusion
  Progression-free survival (PFS) was defined as the time from initiation of IASO104 injection treatment to disease progression or death from any cause, whichever occurred first.
Overall Survival (OS) | Minimum 2 years after IASO104 infusion
  Overall survival (OS) was defined as the time from initiation of IASO104 injection treatment to death from any cause.
Time to Response (TTR) | Minimum 2 years after IASO104 infusion
  Time to response (TTR) was defined as the interval from initiation of IASO104 injection treatment to first achievement of disease response (≥ partial response [PR]).
Time to Complete Response (TTCR) | Minimum 2 years after IASO104 infusion
  Time to complete response (TTCR) was defined as the interval from initiation of IASO104 injection treatment to first achievement of complete response (CR) or better (including stringent complete response [sCR])
Minimal Residual Disease (MRD)-negative rate | Minimum 2 years after IASO104 infusion
  Proportion of subjects achieving bone marrow minimal residual disease (MRD)-negativity by next-generation flow cytometry (NGF) following study treatment
Duration of MRD Negativity | Minimum 2 years after IASO104 infusion
  Duration of MRD negativity was defined as the time from first achievement of MRD-negative status to first MRD recurrence (conversion to positive)
Pharmacokinetic (PK) Endpoints | Minimum 2 years after IASO104 infusion
  Peak concentration (C<sub>max</sub>) of CAR-T cells
  Area under the curve (AUC) over:
  0-28 days post-infusion (AUC<sub>0-28d</sub>) 0-90 days post-infusion (AUC<sub>0-90d</sub>) 0-180 days post-infusion (AUC<sub>0-180d</sub>) Infusion to last measurable timepoint (AUC<sub>0-last</sub>)
Pharmacokinetic (PK) Endpoints | Minimum 2 years after IASO104 infusion
  vector copy number (VCN) in peripheral blood Time to peak concentration (T<sub>max</sub>)
  Area under the curve (AUC) over:
  0-28 days post-infusion (AUC<sub>0-28d</sub>) 0-90 days post-infusion (AUC<sub>0-90d</sub>) 0-180 days post-infusion (AUC<sub>0-180d</sub>) Infusion to last measurable timepoint (AUC<sub>0-last</sub>)
Pharmacodynamic (PD) Endpoints | Minimum 2 years after IASO104 infusion
  Levels of soluble BCMA (sBCMA) in peripheral blood at each timepoint
Pharmacodynamic (PD) Endpoints | Minimum 2 years after IASO104 infusion
  concentrations of CAR-T-related inflammatory biomarkers (including CRP, IL-6, and ferritin)

IPD SHARING:
Plan to Share IPD: No